CLINICAL TRIAL: NCT03454425
Title: A Prospective, Randomized, Sham Controlled Study to Evaluate the Safety and Efficacy of ExAblate Subthalomotomy for the Treatment of Parkinson's Disease Motor Features
Brief Title: A Study to Evaluate the Safety and Efficacy of ExAblate Subthalomotomy for the Treatment of Parkinson's Disease Motor Features
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PD010
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; ExAblate; MRgFUS; Sub-Thalamotomy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exablate Subthalamotomy (Experimental): Exablate treatment for Parkinson's Disease Motor Features
  Interventions: Device: Exablate Subthalamotomy
- Sham ExAblate Subthalamotomy (Sham Comparator)
  Interventions: Device: Sham Exablate Subthalamotomy

INTERVENTIONS:
Device: Exablate Subthalamotomy — ExAblate Subthalomotomy for the Treatment of Parkinson's Disease Motor Features
  Other Names: MRgFUS; Subthalamotomy
  Arms: Exablate Subthalamotomy
Device: Sham Exablate Subthalamotomy — Sham ExAblate Subthalomotomy for the Treatment of Parkinson's Disease Motor Features
  Arms: Sham ExAblate Subthalamotomy

SUMMARY:
The objective of this study is to test the efficacy and safety of unilateral subthalamotomy performed using the ExAblate System for the treatment of Parkinson's disease (PD) motor features.

DETAILED DESCRIPTION:
A Prospective, Randomized, Sham Controlled Study to Evaluate the Safety and Efficacy of ExAblate Subthalomotomy for the treatment of Parkinson's disease motor features.

The objective of this prospective, randomized, double-blind (to subjects, examining neurologists and external video-based examination by Movement Disorders neurologist), two-arm study (ExAblate treated arm Vs ExAblate Sham treated control arm) is to confirm the efficacy of ExAblate Model 4000 Type 1 System for the treatment of Parkinson's disease (PD) motor features and to further demonstrate safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 30 years or older
2. Subjects who are able and willing to give consent and able to attend all study visits.
3. Subjects with a diagnosis of PD by UK Brain Bank Criteria as confirmed by a movement disorder neurologist at the site.
4. Predominant motor features/disability from one side of the body (i.e asymmetry index > 1.5) as determined by a movement disorders neurologist.
5. Motor clinical features non-optimally controlled by an adequate medical treatment prescription. An adequate medication prescription is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
6. No major changes in pharmacological regime for PD should be done for the 30 days prior to procedure.
7. Topographic coordinates of the subthalamic nucleus are localizable on MRI so that it can be targeted by the ExAblate device.
8. Able to communicate sensations during the ExAblate MRgFUS treatment Inclusion and exclusion criteria have been agreed upon by two members of the medical team

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the MDS-UPDRS.
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA) or Mattis Dementia Rating Scale of 120 or lower.
7. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
8. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory.
9. Legal incapacity or limited legal capacity as determined by the neuropsychologist
10. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one
11. Subjects with unstable cardiac status including
12. Severe hypertension (diastolic BP > 100 on medication).
13. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy.
14. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
15. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
16. Patient with severely impaired renal function with estimated glomerular filtration rate <30mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis;
17. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
18. Significant claustrophobia that cannot be managed with mild medication.
19. Subject who weight more than the upper weight limit of the MR table and who cannot fit into the MR scanner
20. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
21. History of intracranial hemorrhage
22. History of multiple strokes, or a stroke within past 6 months
23. Subjects with a history of seizures within the past year
24. Subjects with malignant brain tumors
25. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
26. Any illness that in the investigator's opinion preclude participation in this study.
27. Subjects unable to communicate with the investigator and staff.
28. Pregnancy or lactation.
29. Subjects who have an Overall Skull Density Ratio lower than 0.35 as calculated from the screening CT.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Efficacy - MDS-UPDRS | Baseline to 4 months post treatment
  between-group differences in the mean change (from baseline to 4 months) in the motor MDS-UPDRS score for the side contralateral to subthalamotomy (in the treated group) as compared with mean change in the MDS-UPDRS score for the side contralateral to the alleged subthalamotomy (in the sham-procedure group) in the off-medication condition
Safety - Adverse Events | Baseline to 4 Months post treatment
  To evaluate the incidence and severity of adverse events (AE/AEs) associated with ExAblate subthalamotomy for the treatment of PD motor features.

SECONDARY OUTCOMES:
MDS-UPDRS III ON-medication | Baseline to Month 4 post treatment
  MDS-UPDRS III score in the contralateral body side ON-medication condition as measured by the BLINDED assessor
MDS-UPDRS III OFF-medication | Baseline to Month 4 post treatment
  MDS-UPDRS III score in the contralateral body side OFF-medication condition as measured by the UNBLINDED assessor
MDS-UPDRS III- Contralateral ON-medication | Baseline to Month 4 post treatment
  MDS-UPDRS III score in the contralateral body side ON-medication condition as measured by the UNBLINDED assessor
MDS-UPDRS III | Baseline to Month 4 post treatment
  Specific PD motor features sub-scores (rigidity, bradykinesia, tremor) of MDS- UPDRS III in the contralateral body side by visit for the following: OFF and ON-medication condition as measured by the BLINDED assessor
MDS-UPDRS II | Baseline to Month 4 post treatment
  Total score of MDS-UPDRS II
MDS-UPDRS III Blinded assessor | Baseline to Month 4 post treatment
  Total score of MDS-UPDRS III as measured by the BLINDED assessor OFF- and ON-medication
MDS-UPDRS IV | Baseline to Month 4 post treatment
  Total score of MDS-UPDRS IV and separated by each type of motor complication
PDG39 | Baseline to Month 12 post treatment
  Quality of life assessment with the PDQ39.
GIC | Baseline to Month 4 post treatment
  Patient global impression of change from Baseline to Month 4 FU.
Levodopa | Baseline to Month 12 post treatment
  Levodopa equivalent medication change usage (mg).
MDS-UPDRS | Baseline to Month 12 post treatment
  Durability of the reduction in the contralateral motor MDS-UPDRS at 12 months in the treated group (measured only by the UNBLINDED assessor)
MDS-UPDRS | Baseline to Month 12 post treatment
  Change in the total MDS-UPDRS III according to disease severity at baseline (as defined by the MDS-UPDRS III score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario HM Puerta Del Sur. CINAC, Móstoles, Madrid, Spain

REFERENCES:
- [Derived] Martinez-Fernandez R, Natera-Villalba E, Manez Miro JU, Rodriguez-Rojas R, Marta Del Alamo M, Pineda-Pardo JA, Ammann C, Obeso I, Mata-Marin D, Hernandez-Fernandez F, Gasca-Salas C, Matarazzo M, Alonso-Frech F, Obeso JA. Prospective Long-term Follow-up of Focused Ultrasound Unilateral Subthalamotomy for Parkinson Disease. Neurology. 2023 Mar 28;100(13):e1395-e1405. doi: 10.1212/WNL.0000000000206771. Epub 2023 Jan 11. PMID 36631272
- [Derived] Rodriguez-Rojas R, Pineda-Pardo JA, Manez-Miro J, Sanchez-Turel A, Martinez-Fernandez R, Del Alamo M, DeLong M, Obeso JA. Functional Topography of the Human Subthalamic Nucleus: Relevance for Subthalamotomy in Parkinson's Disease. Mov Disord. 2022 Feb;37(2):279-290. doi: 10.1002/mds.28862. Epub 2021 Dec 3. PMID 34859498
- [Derived] Martinez-Fernandez R, Manez-Miro JU, Rodriguez-Rojas R, Del Alamo M, Shah BB, Hernandez-Fernandez F, Pineda-Pardo JA, Monje MHG, Fernandez-Rodriguez B, Sperling SA, Mata-Marin D, Guida P, Alonso-Frech F, Obeso I, Gasca-Salas C, Vela-Desojo L, Elias WJ, Obeso JA. Randomized Trial of Focused Ultrasound Subthalamotomy for Parkinson's Disease. N Engl J Med. 2020 Dec 24;383(26):2501-2513. doi: 10.1056/NEJMoa2016311. PMID 33369354